CLINICAL TRIAL: NCT00828360
Title: Efficacy Of Low-Dose Dobutamine Stress-Echocardiography To Predict Cardiac Resynchronization Therapy Response
Brief Title: Dobutamine Stress Echocardiography in Cardiac Resynchronization Therapy (CRT) Patients Selection
Acronym: LODO-CRT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ospedale Santa Maria di Loreto Mare (Other)
Responsible Party: Dr. Carmine Muto, Ospedale Santa Maria di Loreto Mare Napoli
Other Study IDs: LM-001
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Last update posted 2009-01-23 (Estimated); Status verified 2009-01

CONDITIONS: Heart Failure
Keywords: Heart Failure; CRT; Dobutamine echocardiography
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
While cardiac resynchronization therapy (CRT) has a well demonstrated therapeutic effect in selected patients with advanced heart failure (HF) on optimized drug therapy, non-responder rate remains high. The low-dose dobutamine stress-echo (DSE) test to predict positive response to CRT (LODO-CRT) trial is designed to improve patient selection for CRT.

DETAILED DESCRIPTION:
LODO-CRT is a multicenter prospective study enrolling HF patients with conventional indication to CRT (symptomatic stable NYHA class III-IV on optimized drug therapy, QRS≥120 msec, left ventricular (LV) dilatation, LVEF≤35%) is designed to assess the predictive value of LV contractile reserve (LVCR), determined through DSE, in predicting CRT response during follow-up. Assessment of CRT effects will follow two sequential phases: in phase 1 CRT response end-point is defined as left ventricular end-systolic volume (LVESV) reduction ≥ 10% at 6 months; in phase 2, both LVESV reduction and clinical status via a clinical composite score will be evaluated at 12 months follow-up. Predictive value of LVCR will be compared to other measures, such as LV dyssynchrony measures, through adjusted multivariable analysis. For the purpose of the study, target patient number is 270 patients (with 95% confidence, 80% power, α≤0.05).

LVCR assessment, using low-dose DES test, should effectively predict positive response to CRT both in terms of the reverse remodeling process as well as favorable long-term clinical outcome. Moreover, the predictive value of LVCR will be compared to that of conventional intra-LV dyssynchrony measures.

ELIGIBILITY:
Inclusion Criteria:

* severe HF despite optimized medical therapy
* NYHA functional class III-IV
* dilated cardiomyopathy of both ischemic and non-ischemic origin
* left ventricular ejection fraction (LVEF) <=35%
* QRS complex duration ≥120 ms
* normal sinus rhythm.

Exclusion Criteria:

* younger than 18 years old
* unstable angina
* acute myocardial infarction
* coronary artery bypass graft (CABG) or percutaneous transluminal coronary angioplasty (PTCA) within the past 3 months
* already implanted with a conventional implantable pulse generator or with an implantable cardioverter defibrillator (ICD)
* previously implanted with a CRT device
* chronic permanent atrial arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient indicated to CRT according to current guidelines
Sampling Method: Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2006-07; Primary Completion 2009-04 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients showing left ventricular reverse remodelling. In particular, a 10% or greater reduction of the left ventricular end-systolic volume (LVESV) is the primary endpoint of the LODO-CRT study. | 6 months

SECONDARY OUTCOMES:
Clinical composite score, which combines changes in the NYHA class and global assessment with the information provided from the occurrence of major clinical events. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Carmine Muto, MD, Principal Investigator — Ospedale Santa Maria di Loreto Mare Naples
Locations (5):
- Italy (5):
  - Anthea Clinic, Bari
  - Sant'Anna Hospital, Catanzaro
  - Istituto Clinico Humanitas, Milan
  - Ospedale Santa Maria di Loreto Mare, Naples
  - Santa Maria della Misericordia, Rovigo

REFERENCES:
- [Background] Muto C, Gasparini M, Iacopino S, Peraldo C, Curnis A, Sassone B, Diotallevi P, Davinelli M, Valsecchi S, Tuccillo B. Efficacy of LOw-dose DObutamine stress-echocardiography to predict cardiac resynchronization therapy response (LODO-CRT) multicenter prospective study: design and rationale. Am Heart J. 2008 Oct;156(4):656-61. doi: 10.1016/j.ahj.2008.06.011. Epub 2008 Aug 27. PMID 18926147